CLINICAL TRIAL: NCT01410513
Title: A Phase 1b, Multicenter, Open-Label, Dose Escalation Study of SAR245409 to Evaluate the Safety, Tolerability and Clinical Activity of SAR245409 in Combination With Rituximab or Bendamustine Plus Rituximab in Patients With Relapsed or Refractory Indolent B-cell Non-Hodgkin Lymphoma, Mantle Cell Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Study Combining SAR245409 With Rituximab or Bendamustine Plus Rituximab in Patients With Indolent Lymphoma, Mantle Cell Lymphoma and Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD12012; U1111-1119-2906 (Other: UTN)
Record Dates: First submitted 2011-07-26; First posted 2011-08-05 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2014-09

CONDITIONS: Indolent Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — XL765

ARMS (3):
- SAR245409 + rituximab (Experimental): Subjects will receive oral SAR245409 twice daily continuously and weekly rituximab intravenously
  Interventions: Drug: SAR245409
- SAR245409 + rituximab + bendamustine (iNHL, MCL) (Experimental): Subjects will receive oral SAR245409 twice daily continuously and monthly bendamustine intravenously.
  Interventions: Drug: SAR245409
- SAR245409 + rituximab+ bendamustine (CLL) (Experimental): Subjects will receive oral SAR245409 twice daily continuously and monthly bendamustine and rituximab intravenously
  Interventions: Drug: SAR245409

INTERVENTIONS:
Drug: SAR245409 — Pharmaceutical form:capsule Route of administration: oral

SUMMARY:
Primary Objective:

- To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for SAR245409 when administered in combination with rituximab or bendamustine plus rituximab

Secondary Objectives:

* To determine the safety and tolerability of SAR245409 in combination with rituximab or bendamustine plus rituximab in subjects with indolent Hon-Hodgkin Lymphoma (iNHL) Mantle Cell Lymphoma (MCL) or Chronic Lymphocytic Leukemia (CLL)
* To determine the pharmacokinetics (PK) of SAR245409, bendamustine and rituximab when used in combination in subjects with iNHL, MCL or CLL
* To determine the pharmacodynamic (PD) effects of SAR245409 in combination with rituximab or bendamustine plus rituximab in subjects with iNHL, MCL or CLL
* To determine the antitumor activity of SAR245409 in combination with rituximab or bendamustine plus rituximab in subjects with iNHL, MCL or CLL

DETAILED DESCRIPTION:
All subjects will take SAR245409 twice daily. All subjects will receive SAR245409 as long as there is clinical benefit.

Combination therapy with SAR245409, bendamustine and rituximab , will be administered over a 28 day cycle for up to 6 to 8 cycles.

Subjects receiving the doublet combination , SAR245409 plus rituximab will receive weekly rituximab for 4 - 8 weeks. Monthly Rituximab may be continued beyond 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* A confirmed diagnosis of indolent non-Hodgkin lymphoma, mantle cell lymphoma or chronic lymphocytic leukemia
* Evaluable disease or measurable disease
* Transfusion independent
* Able to take oral medication
* Male and Female subjects > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Women of childbearing potential using adequate contraception

Exclusion criteria:

* Prior therapy with a PI3K, mTOR or dual PI3K/mTOR inhibitor resulting in adverse events necessitating treatment discontinuation
* Eligible for a hematopoietic stem cell transplant (HSCT)
* The subject has received investigational or non-investigational cytotoxic chemotherapy (i.e., cyclophosphamide), small molecule cancer therapy (i.e., imatinib), biologic cancer therapies other than rituximab (i.e., alemtuzumab, cytokines, vaccines or other monoclonal antibodies) hormonal therapy, radio- or immuno- conjugates (e.g. ibritumomab tiuxetan, tositumomab) or immunosuppressants to treat malignancy within 4 weeks prior to Cycle 1, Day 1
* Radiation therapy within 2 weeks prior to Cycle 1, Day 1
* Autologous Hematopoietic Stem Cell Transplant (HSCT) within the past 16 weeks
* Prior allogeneic HSCT
* Active central nervous system (CNS) metastases or leptomeningeal involvement
* Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C Antibody (anti-HCV)
* Hereditary or acquired immunodeficiency syndrome or human immunodeficiency virus (HIV) infection
* Active peptic ulcer disease requiring treatment with proton pump inhibitors (e.g. pantoprazole) or Type 2 histamine antagonists (e.g. cimetidine)
* Diagnosis or treatment for another malignancy within 3 years of enrollment with the exception of complete resection of basal cell or squamous cell carcinoma of the skin, an in situ malignancy or low-risk prostate cancer after curative therapy
* Inadequate bone marrow function
* Abnormal liver function
* Abnormal renal function
* Abnormal coagulation

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Identification Of Dose-Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) | 4 weeks to 8 weeks

SECONDARY OUTCOMES:
Number of subjects with treatment emergent adverse events | Time from receiving first dose of SAR245409 until 30 days after the last dose
Pharmacokinetics (Cmax) of SAR245409 | up to 2 months
Pharmacokinetics (tmax) of SAR245409 | up to 2 months
Pharmacokinetics (AUC0-12h) of SAR245409 | up to 2 months
Pharmacokinetics (Ctrough) of SAR245409 | up to 2 months
Pharmacokinetics (AUC) of bendamustine | up to 2 months
Pharmacokinetics (AUClast) of bendamustine | up to 2 months
Pharmacokinetics (Ceoi) of bendamustine | up to 2 months
Pharmacokinetics (tmax) of bendamustine | up to 2 months
Pharmacokinetics (Cl) of bendamustine | up to 2 months
Pharmacokinetics (Vss) of bendamustine | up to 2 months
Pharmacokinetics (AUC0-7h) of rituximab | up to 2 months
Pharmacokinetics (Ceoi) of rituximab | up to 2 months
Pharmacokinetics (tmax) of rituximab | up to 2 months
Efficacy as determined by objective response rate (ORR) | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840004, Aurora, Colorado
  - Investigational Site Number 840006, Augusta, Georgia
  - Investigational Site Number 840002, Charleston, South Carolina